CLINICAL TRIAL: NCT06313814
Title: The Effect of Ginger on Functional Dyspepsia Symptoms and Body Fat Content Among Patients With Functional Dyspepsia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Lemlem Gebremariam Aregawi, Principal Investigator, University of Debrecen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DE RKEB/IKEB 5622-2020
Record Dates: First submitted 2024-02-21; First posted 2024-03-15 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- before and after result comparison (Other): we will see if there is an effect after the intervention. we will measure the before and after signs.
  Interventions: Dietary Supplement: Swanson ginger capsule

INTERVENTIONS:
Dietary Supplement: Swanson ginger capsule — Swanson Ginger Root? gingerols, shogaols, and paradols, and possesses multiple bioactivities, such as antioxidant, anti-inflammatory, and antimicrobial properties.
  Ginger is most commonly associated as a culinary spice flavouring to oriental dishes and even the local bakery character biscuit, the gingerbread man. But since ancient times the spice has also been recognized for its health properties, most popular being to settle the stomach, alleviate indigestion and event prevent motion sickness. More recently research has confirmed Ginger's historical effectiveness on digestive health and beyond.

SUMMARY:
The goal of this clinical trial is to assess ginger's effect on patients with functional dyspepsia.

The main question[s] it aims to answer are:

1. Does ginger intake improve functional dyspepsia symptoms?
2. Does ginger intake decrease the body fat content among patients with functional dyspepsia? Dyspepsia patients will be asked to take 540 mg of ginger capsule twice a day. Researchers will assess if there is an improvement in the symptoms of the disease and the fat content. [ to see if gingers effect.

DETAILED DESCRIPTION:
Brief description of the study:

Currently, the options for managing functional dyspepsia are limited and far from ideal. Few conducted studies showed that ginger consumption has a therapeutic and preventive effect on functional dyspepsia however, the results were not conclusive. Therefore, this study will try to investigate the effect of ginger supplementation on functional dyspepsia symptoms and body fat content among patients with Functional dyspepsia.

Volunteers with functional dyspepsia 62 participants will be will take as tablets containing 540mg ginger capsule twice a day for four weeks with follow-up. Functional dyspepsia symptoms will be asked before and after the intervention using a questionnaire based on the symptoms of Rome IV criteria, including gastric fullness, early satiety, nausea, vomiting, belching, epigastric pain and heartburn which will be graded through visual analog scales (0- 10 scores) and measured for the body contents.

Method and Materials

Sample size, sample selection:

The study will include 62 volunteers with functional dyspepsia, female and male participants between the ages of 18 and 72 years.

Study design This study is a before-after interventional study of patients with functional dyspepsia who come to internal medicine, at the University of Debrecen.

Initiator of the investigation:

Mrs. Lemlem Gebremariam Aregawi, PhD student in Nutritional sciences Dr. Zoltán Csiki, Supervisor

Executor of the study:

1. Mrs. Lemlem Gebremariam Aregawi, PhD student in Nutritional sciences Doctoral school of pharmacology and pharmacotherapy, University of Debrecen Tel- +36204027611 E-mail: lemgmed@yahoo.com
2. Dr. Zoltán Csiki, Supervisor Gastroenterologist DE Medical and Health Sciences Center Department: Institute of Internal Medicine - III. s. Department of Internal Medicine Email: csikiz@gmail.com

Test site:

University of Debrecen OEC, Institute of Internal Medicine - III. s. Clinic of Internal Medicine

Form and process of the examination:

The examination is performed by a specialist (gastroenterologist) and nutrition student of the Institute of Internal Medicine with the help of section assistants familiar with the in-body measurement to measure body minerals, fat, muscle, water and BMI.

In the case of each person examined, a form is filled in, which is also recorded in electronic form. The results of the physical examination of this participant as well as the measured results will be recorded.

Body composition analyzer (InBody720): Patient requirements to be included: empty stomach, empty bladder, light clothes and no shoes for measurement in the early morning on the body composition analyzer. Patients with a pacemaker or with metal in the body will be excluded from measurement on this instrument.

Dosage: Volunteers will take 540mg of ginger capsule twice a day for four weeks.

Dosage Attached: In a separate dossier for each surveyed consumer, a statement of consent.

Design of the study: before and after the interventional study Study subject: volunteer consumers, men, women (18 - 72 years).

Meals:

Diet intervention- 100% ginger powder ground 540mg capsule twice a day dose will be used: each component is characterized by elevated stability. It is prepared using extraction procedures suitable for ingredients of the health food market. The capsule will be provided free of charge and specifically designed for this study.

All patients will be instructed to take one capsule immediately before starting lunch and dinner. During 30 days before the beginning of the study and the 28 days of intervention treatment, all patients will be asked to avoid the use of prokinetic and antisecretory (H2 receptor inhibitors and proton pump inhibitors) drugs. All patients will be also asked to limit the consumption of alcoholic beverages (less than or equal to two drinks per day).

Study group Study group: 62 FD patients Response variables (Dependent variables)

* functional dyspepsia symptoms
* body contents, muscle, fat, minerals and water

Task details:

* Preparation, recruitment of consumers, and selection of participants.
* Signing of prospectuses and statements of consent.
* Carry out a preliminary examination among the applicants. Before
* Self-completion questionnaire.
* Performing in-body tests
* Evaluation of results.

Data analysis method:

Data will be analyzed using SPSS software, version 23.0 (IBM Corp., Armonk, NY, USA). Results will be reported as mean (SD) and median (IQR). The Wilcoxon signed rank test will be used to assess the differences in GI symptoms before and after ginger supplementation. The difference between the concentrations at the given time points (initial concentration) will be calculated, the statistical procedure being the repeat t-test. If the background variables become inhomogeneous, it may be necessary to include covariates in the statistical analysis, in which case covariance analysis will be used. If the normality of the data is not adequate for the test or a normal data distribution cannot be transformed, the non-parametric test will be used. We will examine whether the measured parameters change significantly. The significance level will be set at P = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Functional dyspepsia symptoms

Exclusion Criteria:

* Patients with relevant gastroesophageal reflux symptoms (retrosternal pain, burning, or regurgitation) as well as patients with clear evidence of irritable bowel syndrome will not be included. Patients under treatment with pharmacological substances that could influence the gastrointestinal system, such as prokinetics, ursodeoxycholic acid (UDCA), nonsteroidal anti-inflammatory drugs (NSAIDs), cholagogues, protonpump inhibitors, and H2 blockers, will be asked to interrupt this treatment for one month before starting the study treatment.

Moreover, patients with a previous diagnosis of cancer or with previous surgery of the upper gastrointestinal tract or of the biliopancreatic system (except for cholecystectomy) and patients with active HP infection or with gastric or duodenal ulcer, as well as pregnant women, will be excluded.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional Dyspepsia Symptom Severity | four weeks
  This study will evaluate and measure the expected improvements in functional dyspepsia symptoms. It will be assessed by the Nepean Dyspepsia Index (NDI) questionnaire, among 62 patients with functional dyspepsia treated with ginger supplementation compared to the baseline, by the end of the four-week intervention. This measure focuses on the reduction in symptoms such as pain, discomfort, bloating, and early satiety. Each item on the Nepean Dyspepsia Index questionnaire is usually scored on a Likert scale, with higher scores representing more severe symptoms or greater impairment. I.e. Higher scores on the Nepean Dyspepsia Index indicate more severe dyspeptic symptoms and a greater impact on quality of life. Lower scores indicate milder symptoms and less impairment in quality of life. Therefore, a reduction in Nepean Dyspepsia Index scores in response to ginger supplementation indicates an improvement in symptoms and quality of life for individuals with dyspepsia.
Body Fat Content Analysis | Four weeks
  Changes in body fat content, which will be assessed before and after four weeks of ginger supplementation using the In-Body 270, a non-invasive device that measures body weight, skeletal muscle mass, body fat, and other health parameters at five body parts using two different frequencies. This measure aims to evaluate the impact of Functional Dyspepsia and ginger supplementation on body composition, which could be relevant due to potential associations between functional dyspepsia and alterations in body fat distribution.

SECONDARY OUTCOMES:
Improvement in Quality of Life | Four weeks
  Improvements in quality of life will be assessed by the EuroQol Group's EQ-5D questionnaire before and after 4 weeks of ginger supplementation. EuroQol Group's EQ-5D consists of 2 main components:
  1. Descriptive System: This part evaluates health status across 5 dimensions:
     Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression Each is rated on a 3-level scale: 1: No problems to 3: Extreme problems
  2. Visual Analog Scale (VAS): Respondents rate on a scale from 0 to 100, where: 0: Represents the worst imaginable health state 100: Represents the best imaginable health state
  The values for EQ-5D ratings are as follows:
  For each dimension in the descriptive system, the minimum value is 1 (indicating no problems) and the maximum value is 3 (indicating extreme problems).
  For the VAS, the minimum value is 0 (worst imaginable health state) and the maximum value is 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Debrecen, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aregawi LG, Zoltan C. Evaluation of Adverse Effects and Tolerability of Dietary Ginger Supplementation in Patients With Functional Dyspepsia. Curr Ther Res Clin Exp. 2025 Apr 14;102:100792. doi: 10.1016/j.curtheres.2025.100792. eCollection 2025. PMID 40474983